CLINICAL TRIAL: NCT04779164
Title: The Relation Between Abdominal Obesity, Type 2 Diabetes Mellitus and Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir City Hospital (Other)
Responsible Party: Principal Investigator, Fulya Bakılan, principal investigator, Eskisehir City Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: EskCityHosp
Record Dates: First submitted 2021-02-25; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; type 2 diabetes
MeSH Terms: conditions — Osteoarthritis, Knee; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Both patients with and without diabetes mellitus was evaluated in terms of pain and ultrasonographic femoral cartilage thickness.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with type 2 diabetes (Experimental): Patients with diabetes mellitus was evaluated in terms of pain scores and ultrasonographic femoral cartilage thickness and retrospective radiographic knee osteoarthritis scores.
  Interventions: Diagnostic Test: knee ultrasonography
- Patients without type 2 diabetes (Other): Patients without diabetes mellitus was evaluated in terms of pain scores and ultrasonographic femoral cartilage thickness and retrospective radiographic knee osteoarthritis scores.
  Interventions: Diagnostic Test: knee ultrasonography

INTERVENTIONS:
Diagnostic Test: knee ultrasonography — The knees of all patients were screened with ultrasonography device for the measurement of femoral cartilage thicknesses.

SUMMARY:
Background:Knee osteoarthritis is more common in patients with type-2 diabetes mellitus, however it is not known whether this effect is caused by diabetes itself or concominant abdominal obesity.

Objectives:The aim of this study is to determine whether type-2 diabetes itself, independent of abdominal obesity, is a risk factor for femoral cartilage, knee osteoarthritis and poor quality of life.

Design:A cross-sectional design. Settings:Training and research hospital in Turkey. Patients and Methods:Female patients was enrolled in this study and divided into two groups: according to presence or absence of diabetes. Later, both the patients with and without abdominal obesity was divided into two groups according the presence of diabetes.

Main Outcome measures:Clinical parameters were visual analog-scale, gait speed and short form-36. Knee radiographs were evaluated according to Kellgren Lawrance-Scale. And ultrasonography parameters were the measurements of distal femoral cartilage thickness.

Sample size:126

ELIGIBILITY:
Inclusion Criteria:

* being female
* aged between 40 and 70.

Exclusion Criteria:

* Patients with any concomitant chronic disease
* rheumatoid arthritis
* cardiac diseases (except type 2 diabetes mellitus and hypertension)
* knee surgery
* trauma
* bone mass or cancer
* inflammatory arthritis
* impaired cognitive status
* immobilized patients
* type 1 diabetes mellitus

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Knee osteoarthritis is more common in women.
Enrollment: 126 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Femoral cartilage thickness | baseline
  Measured by ultrasonography (higher value:thick cartilage, lower value:thin cartilage)

SECONDARY OUTCOMES:
visual analog scale | baseline
  pain measurement (point 0 to 10) 0:worse pain 10:no pain
radiographic knee osteoarthritis | baseline
  evaluated by kellgren lawrance scale.(0-4) 0:no osteoarthritis, 4: severe osteoarthritis

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Bakılan, Principal Investigator — Eskisehir City Hospital
Locations (1):
- Eskişehir City Hospital, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
1 year later